CLINICAL TRIAL: NCT02565446
Title: Transforming Non-Invasive Liver Disease Detection by MRE: The Hepatogram
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Alina M. Allen, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-003148; K23DK115594 (NIH)
Record Dates: First submitted 2015-09-24; First posted 2015-10-01 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Fatty Liver
MeSH Terms: conditions — Obesity; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric (Experimental): Obese adult subjects who are scheduled to undergo bariatric surgery
  Interventions: Procedure: Magnetic Resolution Elastography (MRE)
- Clinical (Experimental): Subjects who received abdominal surgery for non-liver related indications (cholecystectomy, pancreatic cyst resection)
  Interventions: Procedure: Magnetic Resolution Elastography (MRE)

INTERVENTIONS:
Procedure: Magnetic Resolution Elastography (MRE) — Magnetic Resolution Elastography (MRE): Three-dimensional magnetic resonance elastography (3DMRE), Waves at frequencies of 30 Hz, 40 Hz, and 60 Hz.

SUMMARY:
A variety of liver insults lead to pathological changes in liver architecture that culminate in cirrhosis. While invasive liver biopsy was required to detect cirrhosis, the development of magnetic resonance elastography (MRE) has revolutionized our ability to detect liver fibrosis through non-invasive means that involve measurement of liver stiffness. However, a number of pathological findings occur in liver in response to various insults that precede cirrhosis and are clinically important to identify such as steatosis associated with NASH, inflammation associated with viral hepatitis, and congestion associated with cardiac hepatopathy. Detection of such entities provides essential diagnostic, prognostic, and treatment information but yet is not available non-invasively. Recent murine studies from this group of investigators has identified that MRE technology can be adapted to non-invasively detect these conditions. Implementing this into the practice will transform it by obviating the need for invasive liver biopsies in patients suspected of having such forms of suspected liver disease. This will differentiate Mayo from other institutions where such technology is not available.

An additional aim of this study is to examine the impact of obstructive sleep apnea (OSA) on the pathogenesis of nonalcoholic fatty liver disease (NAFLD), both common comorbidities of obesity. Recent evidence indicates a potential link between OSA and severity of NASH and fibrosis, but the mechanisms of OSA- associated hypoxia on liver disease progression in NAFLD is unclear. This study offers the unique opportunity to analyze this association, as the study population will undergo routine evaluation for OSA, as part as the preoperative work-up prior to bariatric surgery.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age ≥ 18 years
2. Verbal and written fluency of the English Language
3. Able to consent

EXCLUSION CRITERIA

1. Absolute contraindications to MRI including pacemaker, automatic implantable cardioverter/defibrillator (AICD) device, cochlear implant, ventriculoperitoneal (VP) shunt, aneurysm clip, deep brain stimulator, and severe claustrophobia
2. Absolute contraindications to liver biopsy including coagulopathy
3. History of decompensated cirrhosis complicated by one or more of the following: esophageal variceal hemorrhage, ascites, hepatic encephalopathy, or spontaneous bacterial peritonitis.
4. Women who are pregnant or breastfeeding
5. History of liver transplantation or hepatic resection
6. History of primary or secondary hepatic malignancy
7. Current or previous excessive alcohol consumption within 6 months of study enrollment defined as > 30 grams/day for men and > 20 grams/day for women
8. Current or prior history of therapy for underlying liver disease including interferon-based medications, other antiviral agents, immunomodulatory therapy, biologic response modifier therapy, and complementary/alternative medications including (but not encompassing) milk thistle
9. Any severe medical condition that, in the opinion of the Principal Investigator, would serve as an exclusion criterion for study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2015-09; Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
The role of MRE as a non-invasive tool for estimation of inflammation and fibrosis in NAFLD. | The outcome (correlation of liver histology with MR elastogram) will be assessed once, at the time of outpatient biopsy, then again 1 year later with a second biopsy and a second MRE. Outcomes will be assessed after second biopsy.
  120 participants evaluated at Mayo clinic with a diagnoses of NAFLD who are at risk to have NASH. All subjects will undergo an MRE and outpatient liver biopsy.The liver tissue will be assessed for fat, inflammation, and fibrosis by pathology. We are looking for differentiation of simple steatosis from steatohepatitis and steatohepatitis with fibrosis by non-invasive measures such as MRE.

CONTACTS AND LOCATIONS:
Overall Officials: Alina Allen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Wu H, Zhu Z, Li J, Qiu C, Xu P, Glaser KJ, Murphy MC, Venkatesh SK, Yaqoob U, Graham R, Mounajjed T, Manduca A, Winkelmann CT, Yashiro H, Manohar R, Allen AM, Shah VH, Ehman RL, Yin M. Three-Dimensional Vector MR Elastography for Evaluating Tissue Mechanical Heterogeneity to Assess Liver Disease Progression. Radiology. 2025 Apr;315(1):e242349. doi: 10.1148/radiol.242349. PMID 40167439
- [Derived] Li J, Lu X, Zhu Z, Kalutkiewicz KJ, Mounajjed T, Therneau TM, Venkatesh SK, Sui Y, Glaser KJ, Hoodeshenas S, Manduca A, Shah VH, Ehman RL, Allen AM, Yin M. Head-to-head comparison of magnetic resonance elastography-based liver stiffness, fat fraction, and T1 relaxation time in identifying at-risk NASH. Hepatology. 2023 Oct 1;78(4):1200-1208. doi: 10.1097/HEP.0000000000000417. Epub 2023 May 1. PMID 37080558
- [Derived] Allen AM, Shah VH, Therneau TM, Venkatesh SK, Mounajjed T, Larson JJ, Mara KC, Schulte PJ, Kellogg TA, Kendrick ML, McKenzie TJ, Greiner SM, Li J, Glaser KJ, Wells ML, Chen J, Ehman RL, Yin M. The Role of Three-Dimensional Magnetic Resonance Elastography in the Diagnosis of Nonalcoholic Steatohepatitis in Obese Patients Undergoing Bariatric Surgery. Hepatology. 2020 Feb;71(2):510-521. doi: 10.1002/hep.30483. Epub 2019 Mar 15. PMID 30582669
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials